CLINICAL TRIAL: NCT07395518
Title: A Randomized Controlled Trial Comparing the Incidence of Surgical Site Infections in Cesarean Section With and Without Subcutaneous Drain Placement at Queen Savang Vadhana Memorial Hospital
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 014/2568
Record Dates: First submitted 2026-01-13; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Surgical Site Infection (SSI)
Keywords: Cesarean section wound infection; Subcutaneous incision drainage; Elective and Emergency Cesarean section wound infection.
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial (RCT) in which participants are divided into two groups:
  Block randomization will be used, employing a block size of four to ensure a balanced number of participants in both groups.
  Intervention Group: Pregnant women undergoing cesarean section with placement of a subcutaneous wound drain.
  Control Group: Pregnant women undergoing cesarean section without placement of a subcutaneous wound drain.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pregnant women undergoing cesarean section with placement of a subcutaneous wound drain.
  Interventions: Device: Radivac drain
- Control group (No Intervention): Pregnant women undergoing cesarean section without placement of a subcutaneous wound drain.

INTERVENTIONS:
Device: Radivac drain — In the intervention group, a subcutaneous wound drain is placed using a closed suction Redivac drain (10-14 French). The drain is inserted into the subcutaneous layer above the surgical incision through a skin exit site located 2-3 cm from the wound edge, avoiding visible vessels to reduce bleeding. A trocar is used to guide placement, ensuring the drain lies transversely beneath and covers the entire length of the incision. The drain is secured to the skin with silk sutures, connected to a Redivac suction system to apply negative pressure, and covered with a sterile dressing after skin closure to reduce the risk of contamination.
  Arms: Intervention group

SUMMARY:
To study and compare the incidence of surgical site infection after cesarean section in pregnant women with subcutaneous wound drainage and those without subcutaneous wound drainage at Queen Savang Vadhana Memorial Hospital, Sriracha. Chonburi Thailand

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) designed to compare the incidence of surgical site infection after cesarean section between patients who receive subcutaneous wound drainage (Radivac drain) and those who do not. Postoperative wound follow-up will be conducted on postoperative days 3, 7, and 14.

Participants will be randomly assigned into two groups, with the control group consisting of pregnant women undergoing cesarean section at Queen Savang Vadhana Memorial Hospital, Sriracha. Data will be collected on surgical site infection, pain, postoperative complications, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to communicate in Thai
* Undergoing cesarean section, both elective and emergency procedures
* Subcutaneous fat thickness ≥ 4 cm, measured preoperatively using a standardized ultrasound technique
* Able to return for postpartum follow-up at Somdech Phra Boromrajthevi Hospital, Sriracha
* Willing to participate in the study and able to provide written informed consent

Exclusion Criteria:

* Pregnant women with chronic immunosuppressive conditions, such as systemic lupus erythematosus (SLE), HIV infection, severe anemia (Hb < 10.0 g/dL), or uncontrolled diabetes
* Presence of skin disease or skin infection at the abdominal surgical site
* Evidence of infection prior to cesarean section
* Abnormal bleeding disorders requiring specialized treatment
* History of allergy to, or complications from, the use of wound drainage systems
* Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 86 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 14 days
  To compare the incidence of surgical site infection after cesarean section in pregnant women with and without subcutaneous wound drainage.

SECONDARY OUTCOMES:
Length of hospital stay | 14 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Savang vadhana Memmorial Hospital, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Data was save in form of microsoft excel spreadsheet and SPSS file